CLINICAL TRIAL: NCT06431607
Title: A Phase 2a Randomized, Observer-blind, Dose-finding Study to Evaluate the Immunogenicity and Safety of mRNA-based Multivalent Seasonal Influenza Vaccine Candidates in Adults 18 Years of Age and Older
Brief Title: A Study to Find the Dose and Assess the Immune Response and Safety of a Vaccine Against Influenza in Healthy Younger and Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 222853
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Influenza, Human
Keywords: Influenza; Safety; Reactogenicity; Immunogenicity; mRNA vaccine; Healthy younger adults; Healthy older adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an observer blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (14):
- Flu mRNA_YA_Group 1 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 1
- Flu mRNA_YA_Group 2 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 2
- Flu mRNA_YA_Group 3 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 3
- Flu mRNA_YA_Group 4 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 4
- YA_Active Comparator Group 1 (Active Comparator): Eligible participants receive 1 dose of an active comparator at Day 1 intramuscularly.
  Interventions: Combination Product: Active Comparator 1
- Flu mRNA_OA_Group 1 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 5
- Flu mRNA_OA_Group 2 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 6
- Flu mRNA_OA_Group 3 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 7
- Flu mRNA_OA_Group 4 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 8
- OA_Active Comparator Group 2 (Active Comparator): Eligible participants receive 1 dose of an active comparator at Day 1 intramuscularly.
  Interventions: Combination Product: Active Comparator 2
- Flu mRNA_YA_Group 5 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 9
- YA_Active Comparator Group 3 (Active Comparator): Eligible participants receive 1 dose of an active comparator at Day 1 intramuscularly.
  Interventions: Combination Product: Active Comparator 3
- Flu mRNA_OA_Group 5 (Experimental): Eligible participants receive 1 dose of study intervention at Day 1 intramuscularly.
  Interventions: Biological: Flu Seasonal mRNA Formulation 10
- OA_Active Comparator Group 4 (Active Comparator): Eligible participants receive 1 dose of an active comparator at Day 1 intramuscularly.
  Interventions: Combination Product: Active Comparator 4

INTERVENTIONS:
Biological: Flu Seasonal mRNA Formulation 1 — 1 dose of Flu mRNA Formulation 1 is administered intramuscularly in the non-dominant upper deltoid to YA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_YA_Group 1
Biological: Flu Seasonal mRNA Formulation 2 — 1 dose of Flu mRNA Formulation 2 is administered intramuscularly in the non-dominant upper deltoid to YA at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_YA_Group 2
Biological: Flu Seasonal mRNA Formulation 3 — 1 dose of Flu mRNA Formulation 3 is administered intramuscularly in the non-dominant upper deltoid to YA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_YA_Group 3
Biological: Flu Seasonal mRNA Formulation 4 — 1 dose of Flu mRNA Formulation 4 is administered intramuscularly in the non-dominant upper deltoid to YA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_YA_Group 4
Biological: Flu Seasonal mRNA Formulation 5 — 1 dose of Flu mRNA Formulation 5 is administered intramuscularly in the non-dominant upper deltoid to OA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_OA_Group 1
Biological: Flu Seasonal mRNA Formulation 6 — 1 dose of Flu mRNA Formulation 6 is administered intramuscularly in the non-dominant upper deltoid to OA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_OA_Group 2
Biological: Flu Seasonal mRNA Formulation 7 — 1 dose of Flu mRNA Formulation 7 is administered intramuscularly in the non-dominant upper deltoid to OA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_OA_Group 3
Biological: Flu Seasonal mRNA Formulation 8 — 1 dose of Flu mRNA Formulation 8 is administered intramuscularly in the non-dominant upper deltoid to OA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_OA_Group 4
Combination Product: Active Comparator 1 — 1 dose of active comparator 1 is administered intramuscularly in the non-dominant upper deltoid to YA participants at Day 1.
  Arms: YA_Active Comparator Group 1
Combination Product: Active Comparator 2 — 1 dose of active comparator 2 is administered intramuscularly in the non-dominant upper deltoid to OA participants at Day 1.
  Arms: OA_Active Comparator Group 2
Biological: Flu Seasonal mRNA Formulation 9 — 1 dose of Flu mRNA Formulation 9 is administered intramuscularly in the non-dominant upper deltoid to YA participants at Day 1.
  Other Names: GSK4382276A
  Arms: Flu mRNA_YA_Group 5
Biological: Flu Seasonal mRNA Formulation 10 — 1 dose of Flu mRNA Formulation 10 is administered intramuscularly in the non-dominant upper deltoid to OA participants at Day 1.
  Arms: Flu mRNA_OA_Group 5
Combination Product: Active Comparator 3 — 1 dose of active comparator 3 is administered intramuscularly in the non-dominant upper deltoid to YA participants at Day 1.
  Arms: YA_Active Comparator Group 3
Combination Product: Active Comparator 4 — 1 dose of active comparator 4 is administered intramuscularly in the non-dominant upper deltoid to OA at Day1.
  Arms: OA_Active Comparator Group 4

SUMMARY:
The purpose of this study is to assess the safety and immune response of GlaxoSmithKlines (GSK) messenger RNA (mRNA)-based multivalent vaccine (GSK4382276A) candidate against influenza, administered in healthy younger adults (YA) and older adults (OA).

ELIGIBILITY:
Inclusion Criteria:

1. A male or female between and including 18 and 85 years of age (YAs: 18-64; OAs: 65-85) at the time of the study intervention administration.
2. Healthy participants or medically stable patients as established by medical history and clinical examination. Participants with chronic medical conditions with or without specific treatment (e.g., chronic metabolic, cardiac, pulmonary, renal, hepatic, neurologic, and hematologic diseases) are allowed to participate in this study if considered by the investigator as medically stable. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrolment.
3. Body mass index (BMI) >=18 Kilograms per meter square (kg/m²) and less than or equal to (<=) 35kg/m2.
4. Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits), independently or with the assistance of a caregiver.
5. Written informed consent obtained from the participant prior to performance of any study-specific procedure.
6. Female participants of non-childbearing potential may be enrolled in the clinical study.
7. Female participants of childbearing potential may be enrolled in the clinical study, if the participant:

   * Has practiced adequate contraception for 1 month prior to the study intervention administration, and
   * Has a negative pregnancy test within 24 hours prior to the study intervention administration, and
   * Has agreed to continue adequate contraception for at least 1 month after study intervention administration.

Exclusion Criteria:

1. Participant tested positive for influenza by local health authority-approved testing methods within 180 days prior to Day 1.
2. Current or past malignancy, unless completely resolved without sequelae for greater than (>) 5 years before the study intervention administration (excluding effectively treated basal cell skin cancer).
3. Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing required). HIV-infected individuals may be enrolled if they have been stable on antiretroviral therapy for the past 6 consecutive months, i.e., their treatment has not been modified, their cluster of differentiation 4 (CD4) cell count is >= 200/ cubic millimeter (mm³) and their viral load has been undetectable (i.e., HIV-RNA lesser than (<) 50 copies/milliliter [mL]) (based on medical records, no laboratory testing required).
4. Participants with a history of, or current suspicion of myocarditis, pericarditis, or idiopathic cardiomyopathy (including a history of myocarditis or pericarditis following vaccination with an mRNA COVID-19 vaccine), or presence of any medical condition that increases risk of myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis, eosinophilic granulomatosis with polyangiitis and persistent myocardial infection will be excluded from the study.
5. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention (including polyethylene glycol, egg proteins and aminoglycoside antibiotics).
6. Hypersensitivity to latex.
7. Recurrent history or uncontrolled neurological disorders or seizures, including Guillain-Barré syndrome and Bell's palsy, with the exception of febrile seizures during childhood.
8. Any history of dementia or any medical condition that moderately or severely impairs cognition.
9. Any condition that in the judgment of the investigator would make intramuscular injection unsafe.
10. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the clinical study.
11. Administration of an influenza vaccine within 180 days before enrollment or planned administration prior to Visit 2 (Day 29) after the study intervention administration.
12. Previous vaccination with a mRNA influenza vaccine.
13. Administration of a vaccine not foreseen by the study protocol in the period starting 30 days (Day -30) before the study intervention administration, or planned administration within 28 days (Visit 2 [Day 29]) after the study intervention administration*.

    * If emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced, provided it is used according to the local governmental recommendations and sponsor is notified.
14. Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention during the period beginning 30 days before the study intervention administration, or their planned use during the study period.
15. Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the study intervention administration or planned administration during the study period.
16. Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

    * Up to 3 months prior to the study intervention administration:

    For corticosteroids, this will mean prednisone equivalent >=20 mg/day. Inhaled, intraarticular and topical steroids are allowed.
    * Up to 3 months prior to study intervention administration: long-acting immune-modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies, antitumoral medication.
17. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).
18. Pregnant or lactating female participant.
19. Bedridden participants.
20. Female participant planning to become pregnant or planning to discontinue contraceptive precautions within the 1-month post-dosing period.
21. History of chronic alcohol consumption and/or drug abuse in the past 5 years as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
22. Any study personnel or their immediate dependents, family, or household members.
23. Participants with extensive tattoos covering deltoid region on both arms that would preclude the assessment of local reactogenicity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of antigen 1 antibody | At Day 29
Geometric mean increase (GMI) of Antigen 1 antibody titer | From Day 1 to Day 29
Percentage of participants with antigen 1 seroconversion rate (SCR) | From Day 1 to Day 29
Percentage of participants with antigen 1 titer greater than or equal to (>=) the cut off value at Day 1 | At Day 1
Percentage of participants with antigen 1 titer >= the cut off value at Day 29 | At Day 29

SECONDARY OUTCOMES:
GMT of antigen 2 antibody | At Day 29
GMI of antigen 2 antibody titer | From Day 1 to Day 29
Percentage of participants with Antigen 2 SCR | From Day 1 to Day 29
Percentage of participants reporting each solicited administration site event | Day 1 to Day 7
  The following administration site events are solicited: pain, redness, swelling, lymphadenopathy (defined as localized axillary, cervical or supraclavicular swelling or tenderness ipsilateral to the injection arm).
Percentage of participants reporting each solicited systemic event | Day 1 to Day 7
  The following systemic events are solicited: fever, headache, myalgia, arthralgia, fatigue, chills. Fever is defined as temperature >=38 °C/100.4°F regardless the location of measurement. The route for measuring temperature is oral.
Percentage of participants reporting unsolicited adverse events (AEs) | Day 1 to Day 28
  An unsolicited AE is defined as an AE that is either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow up for solicited events. Unsolicited AEs include both serious and non-serious AEs.
Percentage of participants reporting serious adverse events (SAEs) | Day 1 to Day 183
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, is an abnormal pregnancy outcome, or is a suspected transmission of any infectious agent via an authorized medicinal product.
Percentage of participants reporting adverse events of special interest (AESIs) | Day 1 to Day 183
  The following events are considered as AESI in this study: severe hypersensitivity reactions within 24 hours after study intervention administration, myocarditis/pericarditis and potential immune-mediated diseases (pIMDs).
Percentage of participants reporting medically attended adverse events (MAAEs) | Day 1 to Day 183
  A MAAE is defined as an AE that results in an unscheduled visit to a medical professional (e.g., physicians office visits, emergency room visits or hospitalization).

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/